CLINICAL TRIAL: NCT05673447
Title: An Exploratory Clinical Study of Safety and Efficacy of Anti-CD19 CAR NK Cells in the Treatment of Relapsed/Refractory Diffuse Large B Cell Lymphoma
Brief Title: The Study of Anti-CD19 CAR NK Cells in the Treatment of Relapsed/Refractory Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Nanjing Enricnk Biotech Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2022-251
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-12

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: B-Cell Lymphoma; CD19; CAR-NK; diffuse diffuse large B cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 CAR NK cells (Experimental): CD19-CAR-NK is an allogenic CD19-Targeted chimeric antigen receptor NK-cell (CAR-NK) therapy.
  Interventions: Biological: anti-CD19 CAR NK cells

INTERVENTIONS:
Biological: anti-CD19 CAR NK cells — Patients will receive Fludarabine (30 mg/m2 per day) and Cyclophosphamide (300mg/m2 per day) on day -5, -4, and -3. Doses of 6×10^8, 1×10^9, 1.5×10^9 Anti-CD19 CAR NK cells will infused in each group using the "3 + 3" dose-escalation strategy.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of anti-CD19 CAR NK cells in patients with B-cell Non Hodgkin Lymphoma. 9-12 patients are planned to be enrolled in the dose-escalation trial (6×10^8 cells, 1×10^9 cells, 1.5×10^9 cells). The primary endpoints are DLT, MTD. The secondary endpoints are the overall response rates (ORR) and disease control rate (DCR).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this clinical study and sign the Informed Consent Form (ICF).
2. Clinical diagnosis of CD19 positive diffuse large B cell lymphoma as defined by the 2017 World Health Organization (WHO) classification of tumors of haematopoietic and lymphoid tissue.
3. Relapsed/Refractory diffuse large B cell lymphoma refers to: not complete response (CR) of 2 lines of standard treatment; PD after treatment or duration of SD less than 6 months after treatment; progress or relapse within 12 months after autologous stem cell transplant.
4. Subjects with a measurable or evaluable lesion (more than one lesion≥15mm) according to IWG criteria.
5. Age≥ 18 years old and ≤ 75 years old, male or female.
6. Subjects with estimated survival > 12 weeks.
7. Serum albumin (ALB) ≥30g/L, Total Bilirubin (TBIL) ≤ 25.7μmol/L, serum creatinine (SCr) ≤ 132.6μmol/L, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN).
8. Absolute neutrophil count (ANC) ≥ 1.0×109/L, platelet count ≥ 50×109/L.
9. ECOG performance ≤ 1.
10. Left ventricular ejection fraction (LVEF) ≥50% and no clinically significant pericardial effusion.
11. ≥ 4 weeks after subjects received last dose treatment (Radiotherapy, chemotherapy, monoclonal antibody therapy or other treatments).

Exclusion Criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, tozumabs), or subjects with a history of severe allergic reactions.
2. Relapsed after allogenic haemopoietic stem cell transplantation (HSCT).
3. Subjects with active infection receiving intravenous (IV) antibiotic treatment, or received intravenous (IV) antibiotic treatment within one week prior to anti-CD19 CAR NK Cell infusion.
4. Subjects with acquired and congenital immunodeficiency diseases.
5. Subjects with grade III or IV heart failure (NYHA classification).
6. History of epilepsy or other central nervous system (CNS) diseases.
7. Subjects with extranodal lymphoma in Intracranial, lung, or gastrointestinal tract.
8. History of other primary malignant tumors except:

   1. Cured non-melanoma skin cancer by surgical excision, for example basal cell carcinoma (BCC);
   2. Cured primary malignant tumors, such as cervical cancer, superficial bladder cancer, breast cancer.
9. Systemic corticosteroids are used concomitantly within 2 weeks prior to treatment.
10. Females who are pregnant, lactating, or planning a pregnancy within six months.
11. Subjects who have received other clinical trial treatment within 3 months.
12. Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | within 4 weeks after infusion
  To characterize the safety, tolerability, and determine the Maximum tolerated dose (MTD) of Anti-CD19 CAR NK Cells for Relapsed/Refractory diffuse large B cell lymphoma.
Incidence of Treatment Emergent Adverse Events (TEAEs) | up to 48 weeks after infusion
  To characterize the safety of Anti-CD19 CAR NK Cells for Relapsed/Refractory diffuse large B cell lymphoma

SECONDARY OUTCOMES:
The overall response rate (ORR) | 1, 3, 6 and 12 months after infusion
  To characterize the efficacy of Anti-CD19 CAR NK Cell Therapy for Relapsed/Refractory diffuse large B cell lymphoma
Disease control rate (DCR) | 1, 3, 6, 12 and 12 months after infusion
  To characterize the efficacy of Anti-CD19 CAR NK Cell Therapy for R/R Non-Hodgkin Lymphoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No